CLINICAL TRIAL: NCT04932057
Title: The Investigation of Acute Effects of Action Observation Training on Upper Extremity Functionality, Reaction Time and Cognitive Functions in Right-handed Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Yusuf EMUK, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Izmir Katip Celebi University
Record Dates: First submitted 2021-06-13; First posted 2021-06-18 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Right-handed Healthy Adults
MeSH Terms: interventions — Observation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Self-Action Observation (s-AO Group) (Experimental): Participants will watch their own actions during an upper extremity functionality test.
  Interventions: Other: Action observation Training
- Action Observation (AO Group) (Experimental): Participants will watch a person while performing an upper extremity functionality test.
  Interventions: Other: Action observation Training
- Action Practice (Active Comparator): Participants will perform an upper extremity task 4 more times.
  Interventions: Other: Action Practice
- Observation (Placebo Comparator): Participants will watch a slide show which will only contain landscapes.
  Interventions: Other: Observation
- Control (No Intervention): Participants will wait without any performance till the second assesment.

INTERVENTIONS:
Other: Action observation Training — Action observation training is a relatively new rehabilitation approach in which the subject is asked to carefully observe the actions presented through a video clip or performed by an operator.
  Arms: Action Observation (AO Group); Self-Action Observation (s-AO Group)
Other: Action Practice — Participants perform an upper extremity functionality test a couple of times.
  Arms: Action Practice
Other: Observation — Participants will watch a slide show of landscape
  Arms: Observation

SUMMARY:
The aim of the study is to investigate the acute effects of action observation training on upper extremity functionality, reaction times, and cognitive functions in right-handed healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* willingness

Exclusion Criteria:

* any kind of neurological or musculoskeletal problems
* sight problems
* pain in the upper limb
* left handedness

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in upper extremity functionality | The outcome will be assessed at baseline and immediately after the intervention.
  Jebsen-Taylor Hand Function Test will be used
Change in upper extremity dexterity | The outcome will be assessed at baseline and immediately after the intervention.
  Nine-Hole Peg Test will be used.
Change in cognitive functions | The outcome will be assessed at baseline and immediately after the intervention.
  Serial Reaction Time Task will be used.
Change in cognitive functions | The outcome will be assessed at baseline and immediately after the intervention.
  d2 Test of Attention will be used.
Change in reaction time | The outcome will be assessed at baseline and immediately after the intervention.
  Ruler drop test will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emuk Y, Kahraman T, Sengul Y. The acute effects of action observation training on upper extremity functions, cognitive processes and reaction times: a randomized controlled trial. J Comp Eff Res. 2022 Sep;11(13):987-998. doi: 10.2217/cer-2022-0079. Epub 2022 Jun 30. PMID 35770659